CLINICAL TRIAL: NCT07160647
Title: The Efficacy and Safety of Neoadjuvant Therapy With Iparomlimab and Tuvonralimab in Locally Advanced MSI-H/dMMR Colorectal Cancer: An Prospective, Single-Arm Study (Neo-IT)
Acronym: Neo-IT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Sheng Dai, Vice director, Colorectal Surgery, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH2025-0483
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: dMMR/MSI-H-type Rectal Adenocarcinoma
Keywords: Iparomlimab and Tuvonralimab; MSI-H; dMMR; Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a combined treatment regimen of immunotherapy and radical surgical resection (Experimental): Eligible patients with advanced MSI-H/dMMR colorectal cancer will receive a combined treatment regimen of immunotherapy and radical surgical resection. The specific procedures are as follows:
  Anti-PD-1/CTLA-4 dual immunotherapy (5 mg/kg, IV, D1, Q3W, 4 cycles). Radical surgical resection will be performed after the completion of immunotherapy.
  Interventions: Drug: Ipalolimab and Tovorilimab

INTERVENTIONS:
Drug: Ipalolimab and Tovorilimab — 1.Active Ingredients: Ipalolimab and Tovorilimab (a dual-functional combination antibody consisting of Ipalolimab, a recombinant humanized monoclonal antibody targeting programmed death receptor-1 [PD-1], and Tovorilimab, a recombinant humanized monoclonal antibody targeting cytotoxic T-lymphocyte-associated protein-4 [CTLA-4]). 2.Specification: 50 mg (2 mL) per vial. 3.Dosage and Administration: Administer via intravenous infusion at a recommended dose of 5 mg/kg every 3 weeks.

SUMMARY:
Immunotherapy may bring revolutionary changes to the preoperative neoadjuvant treatment mode for dMMR/MSI-H locally advanced rectal cancer. According to the existing theory, the use of Iparomlimab and Tuvonralimab may be the best solution. In this study, the investigators will perform single-cell sequencing of participants tissue samples, fully explore the multi-dimensional omics information of tumors and microenvironments, explore the characteristics of the treatment benefit population, and try to construct an efficacy prediction model to screen the treatment benefit population early and implement precise treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to receive neoadjuvant therapy.
2. Age ≥18 years.
3. Histologically confirmed primary colorectal adenocarcinoma (without squamous or sarcomatoid components).
4. Radiologically assessed (contrast-enhanced CT or MRI) as surgically resectable stage IIB-III (limited to cT4 or cN+ per AJCC 8th edition).
5. Confirmed dMMR or MSI-H status by immunohistochemistry or MSI genetic testing.
6. Lesions diagnosed by investigators as amenable to radical resection (R0 resection) without requiring multi-organ resection prior to neoadjuvant therapy.
7. Voluntary participation with signed informed consent.
8. ECOG performance status score of 0-1.
9. No prior antitumor or immunotherapy before enrollment.
10. Adequate organ and bone marrow function defined as:

    1. Hematology: Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L; Platelets (PLT) ≥100×10⁹/L; Hemoglobin (HGB) ≥7.0 g/dL.
    2. Liver function: Total Bilirubin (TBIL) ≤1.5×ULN; Alanine Transaminase (ALT) and Aspartate Aminotransferase (AST) ≤3×ULN; Serum Albumin (ALB) ≥28 g/L.
    3. Renal function: Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min; Urine dipstick shows protein <2+; for subjects with baseline urine dipstick protein ≥2+, a 24-hour urine collection must demonstrate protein <1 g.
    4. Coagulation: International Normalized Ratio (INR) ≤1.5 and Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN.
11. No severe comorbidities jeopardizing survival (life expectancy <5 years).
12. Fertile female subjects or male subjects with fertile partners must use effective contraception during and for 6 months after treatment. Postmenopausal status or negative urine/serum pregnancy test for premenopausal females.

Exclusion Criteria:

* 1.Prior antitumor therapy for the disease under investigation, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc.

  2.Previous treatment with anti-PD-1, anti-PD-L1, anti-programmed death ligand 2 (PD-L2), or anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) agents, or any other drugs targeting T-cell co-stimulation or immune checkpoint pathways (e.g., OX40, CD137), as well as adoptive cell immunotherapy.

  3.Concurrent participation in another interventional clinical study. 4.Treatment with any investigational drug or device within 4 weeks prior to the first dose of the study drug.

  5.Within 7 days before screening laboratory tests: receipt of blood transfusion, granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), erythropoietin (EPO), thrombopoietin (TPO), or IL-11 therapy.

  6.Use of immunosuppressive drugs within 4 weeks before the first dose of the study drug, excluding: intranasal/inhaled topical steroids or local steroid injections (e.g., intra-articular); systemic corticosteroids at doses ≤10 mg/day prednisone or equivalent; corticosteroids as premedication for allergic reactions (e.g., CT scan premedication).

  7.Use of Chinese herbal medicine with antitumor indications or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 1 week before the first dose of the study drug.

  8.Receipt of live or attenuated vaccines within 4 weeks before the first dose or anticipated during the study.

  9.Major surgery (e.g., craniotomy, thoracotomy, or laparotomy) within 4 weeks before the first dose, anticipated need for major surgery during the study (except protocol-defined radical resection for colon cancer), or presence of unhealed wounds, ulcers, or fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the pathologic complete response (pCR) rate | Up to 13 weeks (once surgery is done)
  Description: pCR was defined as the absence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes (ypT0N0).

SECONDARY OUTCOMES:
Tumor regression grade | Up to 13 weeks (once surgery is done)
  Tumor Regression Grade（TRG）will be done via pathologic assessment on the surgical specimen with AJCC/CAP TRG system
The proportion of participants who remain survival at 3 years | Up to 3 years
  Defined as the percentage of patients alive after 3-year follow-up
The proportion of participants who remain progression free at 3 years | Up to 3 years
  Defined as the percentage of patients without disease recurrence or progression after 3-year follow-up
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0 | Up to 3 years
  Treatment- related adverse events are assessed by NCI-CTCAE v5.0 in each visit
Quality of life of the patients | up to 3 years
  Quality of life is measured via FACT-C questionnaire in each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Xiujun Cai, MD, Study Chair — Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang 310016
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine,, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided